CLINICAL TRIAL: NCT04475939
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Comparing Niraparib Plus Pembrolizumab Versus Placebo Plus Pembrolizumab as Maintenance Therapy in Participants Whose Disease Has Remained Stable or Responded to First-Line Platinum -Based Chemotherapy With Pembrolizumab for Stage IIIB/IIIC or IV Non-Small Cell Lung Cancer (ZEAL-1L)
Brief Title: Placebo-controlled Study Comparing Niraparib Plus Pembrolizumab Versus Placebo Plus Pembrolizumab as Maintenance Therapy in Participants With Advanced/Metastatic Non-Small Cell Lung Cancer
Acronym: ZEAL-1L
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 213400; 2023-508443-40 (Registry Identifier: CTIS); 2020-002202-20 (EudraCT Number)
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Niraparib; Pembrolizumab; Maintenance therapy; Chemotherapy; Platinum-based
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — niraparib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participant Investigator study staff and the Sponsor study team will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Participants receiving niraparib plus pembrolizumab (Experimental): Eligible participants will receive niraparib along with pembrolizumab.
  Interventions: Drug: Niraparib; Biological: Pembrolizumab
- Participants receiving placebo plus pembrolizumab (Placebo Comparator): Eligible participants will receive matching placebo along with pembrolizumab.
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered.
  Arms: Participants receiving niraparib plus pembrolizumab
Biological: Pembrolizumab — Pembrolizumab will be administered
Drug: Placebo — Matching placebo will be administered
  Arms: Participants receiving placebo plus pembrolizumab

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study of niraparib plus pembrolizumab versus placebo plus pembrolizumab as maintenance therapy in participants with advanced or metastatic non-small cell lung cancer (NSCLC) who have achieved stable disease (SD), partial response (PR), or complete response (CR) following completion of standard of care first-line (SoC 1L) platinum-based induction chemotherapy with pembrolizumab. The primary hypotheses are: participants with confirmed diagnosis of NSCLC could benefit from niraparib plus pembrolizumab versus placebo plus pembrolizumab with respect to Progression-free survival (PFS) and Overall survival (OS).

ELIGIBILITY:
Inclusion criteria:

* Participant must be >=18 years of age.
* Has a histologically or cytologically confirmed diagnosis of NSCLC without known targetable driver alteration (either non-squamous or squamous histology; mixed histology is allowed for which an approved targeted therapy is available in the 1L induction/maintenance therapy setting).
* Has advanced (Stage IIIB or Stage IIIC, not amenable to definitive chemoradiotherapy) or metastatic (Stage IV) or metastatic (Stage IV) NSCLC.
* Has completed at least 4 but no more than 6 cycles of SoC 1L platinum-based induction chemotherapy with pembrolizumab.
* Has SD, PR, or CR of the NSCLC per Investigator's assessment after completion of 4 to 6 cycles of SoC 1L platinum-based induction chemotherapy with pembrolizumab.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a life expectancy of at least 12 weeks.
* Has adequate organ and bone marrow function.
* Must submit tumor specimens.
* Must be able to swallow and retain orally administered study treatment.
* A female is eligible to participate if she is not pregnant or breastfeeding and must follow contraceptive guidance during the treatment period and 180 days afterwards.
* A male is eligible to participate if he agrees to contraceptive guidance and refrains from sperm donation during the intervention period and for at least 90 days after the last dose of study treatment.
* Is able to understand the study procedures and agrees to participate in the study by providing written informed consent. Participants must be informed that their participation is voluntary. Participants will be required to sign a statement of informed consent to participate in the study.

Exclusion criteria:

* Has mixed small cell lung cancer or sarcomatoid variant NSCLC.
* Has received prior Poly (adenosine diphosphate-ribose) polymerase (PARP) inhibitor(s) in prior lines of treatment.
* Has systolic blood pressure (BP) >140 millimeters of mercury (mmHg) or diastolic BP >90 mmHg.
* Has any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* Has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiographic signs of CNS hemorrhage.
* Has received colony-stimulating factors (granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) within 4 weeks prior to the first dose of study treatment.
* Has an active or previously documented autoimmune or inflammatory disorder.
* Is receiving chronic systemic steroids (prednisone >20 mg per day) other than intermittent use of bronchodilators, inhaled steroids, or local steroid.
* Has other active concomitant malignancy that warrants systemic, biologic, or hormonal therapy.
* Is pregnant, breastfeeding, or expecting to conceive children while receiving study treatment and/or for up to 180 days after the last dose of study treatment.
* Has a known history of Myelodysplastic syndrome (MDS) or Acute myeloid leukemia (AML).
* Has a known history of active tuberculosis.
* Has current active pneumonitis within 90 days of planned start of the study or a known history of interstitial lung disease, drug-related pneumonitis, or radiation pneumonitis requiring steroid treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) using Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 in complete and partial response (CR/PR) population | Up to approximately 3 years
  PFS in CR/PR population is defined as the time from the date of randomization to the date of first radiographic progression as determined by BICR or death from any cause in the absence of progression, whichever occurs first.

SECONDARY OUTCOMES:
PFS assessed by BICR using RECIST v 1.1 in intent to treat (ITT) population | Up to approximately 3 years
  PFS in the ITT Population is defined as the time from the date of randomization to the date of first radiographic progression as determined by BICR or death from any cause in the absence of progression, whichever occurs first.
OS in CR/PR population | Up to approximately 3 years
  OS in CR/PR population defined as the time from randomization to the date of death due to any cause.
OS in overall population | Up to approximately 5 years
  OS is defined as the time from randomization to the date of death due to any cause.
Time to progression (TTP) | Up to approximately 3 years
  TTP in the Central nervous system (CNS) is defined as the time from the date of randomization until the earliest date of documented PD in the CNS, based on BICR assessment using response assessment in neuro-oncology brain metastases (RANO-BM) criteria.
PFS by investigator assessment using RECIST v1.1 | Up to approximately 3 years
  PFS is defined as the time from the date of randomization to the date of first radiographic progression as determined by the Investigator using RECIST v1.1 or death from any cause in the absence of progression, whichever occurs first.
CNS PFS as assessed by BICR using RANO-BM | Up to approximately 3 years
  PFS is defined as the time from the date of randomization to the date of first radiographic progression as determined by BICR using RANO-BM criteria or until death due to any cause (whichever occurs first).
PFS as assessed by BICR using RECIST v1.1 by programmed cell death-ligand 1 (PD-L1) status | Up to approximately 3 years
  PFS is defined as the time from the date of randomization to the date of first radiographic progression as determined by BICR using RECIST v1.1 or death from any cause in the absence of progression, whichever occurs first. PFS will be assessed by PD-L1 status (PD-L1 tumor cells [TCs] less than [<]1% and not evaluable (NE) versus more than or equal to [>=]1%).
OS by PD-L1 status | Up to approximately 5 years
  OS is defined as the time from randomization to the date of death due to any cause. OS will be assessed by PD-L1 status (PD-L1-TCs <1% and NE versus >=1%).
Time to Deterioration (TTD) in Lung Symptoms | Up to approximately 3 years
  TTD is defined as the time from randomization to meaningful deterioration as measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire 13-item lung cancer-specific module (EORTC QLQ-LC13) questionnaire
Change from Baseline in Health-related quality of life (HRQoL), functioning and symptoms by EORTC QLQ-C30-item Core module (EORTC QLQ-C30) (Scores on a scale) | Baseline, Day 1 in Cycles 1, 2, 3, 4, 5 (Each cycle is of 21 Days); thereafter every 2 cycles until 90 days after last treatment dose (up to approximately 3 years)
  EORTC QLQ-C30 is a validated questionnaire to assess overall health-related quality of life in participants with cancer.
Change from Baseline in HRQoL functioning and symptoms by EORTC QLQ-LC13 (Scores on a scale) | Baseline, Day 1 in Cycles 1, 2, 3, 4, 5 (Each cycle is of 21 Days); thereafter every 2 cycles until 90 days after last treatment dose (up to approximately 3 years)
  The EORTC QLQ-LC13 is a clinically valid and useful tool for assessing disease- and treatment-specific symptoms in lung cancer participants.
Number of participants with adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | Up to approximately 3 years
  AEs, SAEs and AESIs will be collected.
Plasma concentrations of niraparib | Up to approximately 3 years
  Blood samples will be collected to assess the plasma concentrations of niraparib.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (157):
- United States (22):
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Lone Tree, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Newnan, Georgia
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sherman, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Fairfax, Virginia
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Cipoletti Rio Negro
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Florida
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Rosario
- Australia (4):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Ballarat, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Brazil (7):
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Cachoeiro de Itapemirim
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Uberlândia
- Bulgaria (5):
  - GSK Investigational Site, Panagyurishte
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
- Chile (2):
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Temuco
- Colombia (2):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Montería
- France (10):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Saint-Herblain
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
- Germany (15):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bonn
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Gauting
  - GSK Investigational Site, Großhansdorf
  - GSK Investigational Site, Halle
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Heidelberg
  - GSK Investigational Site, Hemer
  - GSK Investigational Site, Jena
  - GSK Investigational Site, München
  - GSK Investigational Site, Stuttgart
  - GSK Investigational Site, Velbert
- Greece (8):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion Crete
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Neo Faliro
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Pylaia Thessaloniki
  - GSK Investigational Site, Rio Patras
  - GSK Investigational Site, Thessaloniki
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Gyöngyös
  - GSK Investigational Site, Tatabánya
  - GSK Investigational Site, Törökbálint
- Ireland (2):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
- Italy (12):
  - GSK Investigational Site, Avellino
  - GSK Investigational Site, Aviano PN
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Catania
  - GSK Investigational Site, Florence
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Orbassano to
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Verona
- Mexico (3):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
  - GSK Investigational Site, Puebla Puebla
- Netherlands (7):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zwolle
- Norway (3):
  - GSK Investigational Site, Drammen
  - GSK Investigational Site, Lrenskog
  - GSK Investigational Site, Oslo
- GSK Investigational Site, Lima, Peru
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Olsztyn
- Romania (6):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Satu Mare
  - GSK Investigational Site, Timișoara
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
- South Korea (4):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
- Spain (10):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Zaragoza
- Sweden (3):
  - GSK Investigational Site, Gävle
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- GSK Investigational Site, Lausanne, Switzerland
- Turkey (Türkiye) (3):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Edirne
  - GSK Investigational Site, Istanbul
- United Kingdom (5):
  - GSK Investigational Site, Bournemouth
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Middlesex
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Ramalingam SS, Thara E, Awad MM, Dowlati A, Haque B, Stinchcombe TE, Dy GK, Spigel DR, Lu S, Iyer Singh N, Tang Y, Teslenko I, Iannotti N. JASPER: Phase 2 trial of first-line niraparib plus pembrolizumab in patients with advanced non-small cell lung cancer. Cancer. 2022 Jan 1;128(1):65-74. doi: 10.1002/cncr.33885. Epub 2021 Sep 3. PMID 34478166